CLINICAL TRIAL: NCT02092584
Title: Effect of Omega-3 Supplementation on Serum Level and Gene Expression of IGF-1and IGFBP-3 in Men With Cardiovascular Disease.
Brief Title: Effect of Omega-3 Supplementation on Serum Level and Gene Expression of IGF-1and IGFBP-3 in Men With CVD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5144
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Disease
Keywords: atherosclerotic; IGF-1; IGFBP-3
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVD, Omega-3 (Active Comparator): patients with Cardiovascular disease who receive 4g/d omega-3
  Interventions: Dietary Supplement: Omega-3
- CVD, Placebo (Placebo Comparator): patients with cardiovascular disease who receive 4 cap of placebo/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — 4 cap 1 g Omega-3 per day for 2 months
  Other Names: n-3 fatty acids; n-3 PUFA
  Arms: CVD, Omega-3
Dietary Supplement: Placebo — 4 cap 1 g Placebo(paraffin) per day for 2 months
  Arms: CVD, Placebo

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with omega 3 or placebo for 8 weeks in serum level of IGF-1 and IGFBP-3 and gene expression of IGF-1 in patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* CVD patients 45- 65 years old, patients with ≥ 50% stenosis in at least one coronary angiogram demonstrated, body mass index in the range 18.5- 35, avoidance of dietary supplements, vitamins and herbal products at least 3 months before and throughout the intervention, willingness to participation,

Exclusion Criteria:

* people who have used omega 3 supplements in last 3 months, having chronic renal disease , GI disease, hepatobiliary diseases, hematological disorders, hypo- or hyperthyroidism, Smokers

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Serum Total Cholesterol | Change from baseline at 2 months
Serum HDL-C | Change frome baseline at 2 months
Serum LDL-C | Change frome baseline at 2 months
Serum TG | Change frome baseline at 2 months
Serum Fasting Blood Sugar(FBS) | Change frome baseline at 2 months
Serum Insulin | Change frome baseline at 2 months
Serum hsCRP | Change frome baseline at 2 months
Serum Insulin Like Growth Factor-1(IGF-1) | Change frome baseline at 2 months
Serum IGF binding protein 3(IGFBP-3) | Change frome baseline at 2 months

SECONDARY OUTCOMES:
Gene Expression of IGF-1 | Change frome baseline at 2 months
Gene expression of IGFBP3 | change from baseline at 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran